CLINICAL TRIAL: NCT05337020
Title: Survey on the Future of Telemedicine in the Daily Care of Cardiology Patients.
Acronym: MEDICAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-1945
Record Dates: First submitted 2022-03-11; First posted 2022-04-20 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Diseases
Keywords: Telemedicine
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): 240 patients will receive the questionnaire to assess patients vision on telemedicine.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Each patient will be asked to fill in the questionnaire to assess their vision on telemedicine

SUMMARY:
The Cardiology research group at the Jessa Hospital Hasselt and the University Hospital Antwerp (in collaboration with the University of Hasselt and the University of Antwerp) is conducting research into remote patient monitoring (telemedicine). Digital technologies such as smartphones, tablets, fitness trackers, smartwatches,… make it easier to monitor the health of cardio patients between consultations. This would allow for faster intervention when necessary, but consultations can also (partially) take place remotely. For this study, we are looking for patients who have already used such technologies to remotely monitor their health and patients who have never used it before.

We would like to find out how these patients feel about telemedicine by means of a questionnaire. This will take approximately 5 to 10 minutes. In this way, we can gain a better understanding of these patients' views and expectations regarding telemedicine. In this way we can further improve healthcare and develop more options to follow up patients even better from your home environment.

DETAILED DESCRIPTION:
The main aim of this study is to evaluate the overall perception of cardiology patients concerning telemedicine features and services in two patient groups: patients who had already any kind of telemedicine follow-up and a small population which never made us of a telemedicine follow-up.

More specifically the aims are:

* to assess the enablers and barriers to the use of telemedicine.
* to explore the willingness to pay for such telemedicine tools.

This is a multicentric, prospective study performed at Jessa Hospital Hasselt, Belgium and Antwerp University Hospital (UZA), Belgium in which a newly developed questionnaire (Appendix 1) will be used. It takes about 5-10 minutes to fill in the survey. The questionnaire contains 6 parts:

* General information on the patients and the use of telemedicine tools
* Questions about the importance of functions and services in telemedicine tools
* Questions about enablers to use telemedicine
* Questions on the ease-of-use of such technologies
* Questions on barriers using telemedicine
* Questions on the willingness to pay for such telemedicine tools.

Two patient groups will be included: 1. Patients who already had a telemonitoring follow-up in the past and 2. Patients who have never been followed with a telemonitoring tool (except for teleconsultations during COVID-19 without any other telemedicine tools) as a control group. There are at least 2000 patients in Jessa and UZA who have had a form of telemonitoring in the past years (from 2014 untill now): i.e. patients with a cardiovascular implantable electronic device (CIED) followed by the telemonitoring unit, atrial fibrillation patients who received personal follow-up via education or therapy adherence monitoring, patients who received remote heart rhythm monitoring during COVID, patients who participated in telerehabilitation projects and heart failure patients who received intensive telemonitoring via an online platform.

Two recruitment strategies will be applied. Patients who already have had a mHealth follow-up both at Jessa or UZA and are available in a database of the cardiology ward will be approached to participate in this study by phone contact and asked if they want to participate via a link sent via email. If they agree, an email with a link to the questionnaire (Appendix 2) will be sent to these patients. After they approve with the digital informed consent (IFC), they can fill in the questionnaire. Patients who are present at the hospital for an in-person device consultation or hospitalized patients/patients coming for a consultation without a telemonitoring follow-up method in the past will be approached in-person. After a short introduction about the project, the patients will be asked to participate in the study. These patients can approve with the digital IFC after which they can fill in the questionnaire via the tablet in the hospital. A list will be kept of patients who have been approached to avoid patients being asked twice as the questionnaire will be anonymous. In this list, only patients name, first name and patient number will be added. No additional visits are necessary for both recruitment groups. A sample size calculation for this study is not applicable as this is an observational study that includes all eligible patients from mHealth databases available at the cardiology ward or patients coming for an in-person follow-up (at a device consultation)/hospitalized patients. However, the aim is to reach 240 completed forms with at least 40 completed forms in every telemedicine group and the control group. Therefore, specific Qualtrics links will be used for each telemedicine group and a specific link for the control group. This is only for the analyses and sample size. The questionnaire will be the same through all qualtrics links.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a follow-up at the cardiology department of Jessa Hospital Hasselt or UZA
* Participants over the age of 18 years

Exclusion Criteria:

* Participants who are not able to read or fully understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Questionnaire to assess enablers and barriers to use telemedicine | day 1
  to assess the enablers and barriers to the use of telemedicine.
Questionnaire to assess willingness to pay for telemedicine tools | day 1
  to explore the willingness to pay for such telemedicine tools.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Antwerp University hospital, Edegem, Limburg
  - Jessa Hospital Hasselt, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: No